CLINICAL TRIAL: NCT06312241
Title: Feasibility, Acceptance and Efficacy of Metacognitive Training-Silver BeWell in Older Adults
Brief Title: Metacognitive Training-Silver BeWell in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, BViertel, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-Silver BeWell
Record Dates: First submitted 2024-02-19; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Depressive Symptoms; Well-Being, Psychological
Keywords: Metacognitive Training; intervention; older adults; cognitive-behavioral therapy; MCT-Silver
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metacognitive Training-Silver BeWell (Experimental): MCT-Silver BeWell is a cognitive-behavioral therapy based group intervention, which aims to improve insight for and change negative (meta)cognitive beliefs (e.g., negative mental filter), information-processing biases (e.g., mood-congruent memory), unhelpful behaviors (e.g., social withdrawal) and emotion-regulation (ER) strategies (e.g. rumination, avoidance of negative feelings) associated with the onset of depression. The training represents a variant of MCT-Silver for depression in later life developed for older adults without clinical depression.
  Interventions: Behavioral: Metacognitive Training-Silver BeWell

INTERVENTIONS:
Behavioral: Metacognitive Training-Silver BeWell — Metacognitive Training- Silver BeWell is a cognitive behavioral based group intervention, which focuses on helping participants gain (metacognitive) distance from thought and behavioral patterns as well as behaviors and ER-strategies that are implicated in the onset of depression and reduced overall mental well-being. In 10 modules, MCT-Silver addresses issues specific to later life such as coping with physical changes and loss, as well as adapting to new (social) roles. The program also includes modules on identifying and re-defining values in later life, acceptance of negative feelings and resilience. In the training participants are made aware of information processing biases that have been shown to contribute to the onset of depression through engaging exercises using examples from daily life. Groups are comprised of up to 10 participants. Each session is 90 minutes.

SUMMARY:
The present study seeks to examine the feasibility, acceptance and efficacy of Metacognitive Training-Silver (MCT-Silver) BeWell among older adults (ages 60 years and older) delivered in a community setting (e.g., social-psychiatric community center, nursing homes, etc.).

DETAILED DESCRIPTION:
Up to 20% of older adults have major depression and up to 30% have subclinical depressive symptoms (e.g., symptoms of depression that do not fulfill criteria for a major depressive episode). Given that depression in later life is associated with the onset of dementia and disability and that older adults have a higher risk of suicide and a longer time to remission, prompt treatment of subclinical depression and prevention of depression in later life is of importance. However, there is a lack of empirically-based, low-threshold and cost-effective group interventions for older adults, which can be delivered in community settings (e.g., community centers or nursing homes) by community mental health workers.

To fill this gap, the present study seeks to examine the feasibility, acceptance and efficacy of Metacognitive Training-Silver (MCT-Silver) BeWell among older adults (ages 60 years and older) delivered in a community setting (e.g., social-psychiatric community center, nursing homes, etc.). MCT-Silver BeWell is a standardized, cognitive-behavioral therapy based group intervention, which aims to improve insight for and reduce negative (meta)cognitive beliefs (e.g., negative mental filter), unhelpful behaviors (e.g., social withdrawal) and emotion-regulation (ER) strategies (e.g. rumination, avoidance of negative feelings) associated with the onset of depression. Like its forerunners, metacognitive training for psychosis (MCT) and depression in younger and middle-aged adults (D-MCT), MCT-Silver BeWell also aims at correcting information-processing biases (e.g., mood-congruent memory) associated with reduced mood and psychological well-being. In MCT-Silver BeWell sessions, psychoeducation regarding the association between negative (meta)cognitive beliefs and information-processing biases, ER strategies and behaviors with psychological well-being is presented and alternative, more helpful thoughts, strategies and skills are introduced and practiced with the aim of improving overall psychological well-being.

MCT-Silver for depression yielded significant effects beyond an active control group on self-reported depression, rumination and self-reported health in an outpatient setting with older adults with affective disorders, A pilot study of D-MCT among older adults also demonstrated the feasibility of the depression intervention in an inpatient setting and randomized clinical trials of D-MCT with adult sample have demonstrated the short and mid-term efficacy of D-MCT as well as session-specific effects, acceptance and (minimal) side effects.

In the current study, the investigator examine the acceptance, feasibility and efficacy of MCT-Silver BeWell among older adults. The number of sessions attended will serve as the primary outcome. Group attendance is expected to be high. Further outcomes include participants' acceptance (subjective ratings) as well as negative side effects of the intervention. It is expected that participants will rate the intervention positively and will report few negative side effects of the intervention. Other secondary outcomes include depression, resilience, loneliness, self-reported health, dysfunctional beliefs, and rumination

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 60 years or older
* Sufficient command of the German language
* Willingness to participate in intervention over a period of 10 weeks (participants who do not attend the intervention, but complete questionnaires will also be included in the analysis)
* Visual and auditory acuity adequate for participation in group sessions
* Ability to participate in the group setting (ability to participate in the group setting will be assessed during a screening interview (e.g., adequate social skills)).

Exclusion Criteria:

* Acute suicidality as assessed by BDI-II Item 9
* Dementia (MMSE < 24) or evidence of severe organic brain dysfunction

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of sessions attended | 10 weeks (pre (t0)- to post (t1))
  The total number of sessions attended (of 10) will be used to assess the feasibility of the intervention

SECONDARY OUTCOMES:
Participants' appraisal of the training | after each session weeks 1 through 10; post (10 weeks; t1) and follow-up (3 months; t2)
  Participant's acceptance of the training as measured by a self-developed questionnaire; single items assessing patients' acceptance of the training (1 = low acceptance; 5 = high acceptance); high scores indicate better appraisal of the intervention
Negative effects questionnaire (NEQ) | post (10 weeks; t1) and follow-up (3 months; t2)
  Negative effects of the intervention will be assessed by the Negative Effects Questionnaire "negative effects of treatment" score (minimum = 0; maximum = 128); higher scores indicate more negative side effects
Depression (Beck Depression Inventory - II) | baseline (t0), post (10 weeks; t1), and follow-up (3 months; t2)
  Change in self-assessed depression as measured by the Beck Depression Inventory-II (BDI-II) from baseline to post-assessment (t0 to t1) and follow-up (t0 to t2); 21 items are assessed on a 4-point Likert scale; higher scores indicate more depressive symptoms; (minimum score = 0; maximum score = 63)
Dysfunctional beliefs (18-item Dysfunctional Attitudes Scale) | baseline (t0), post (10 weeks; t1), and follow-up (3 months; t2)
  Change in dysfunctional beliefs as measured by the 18-item Dysfunctional Attitude Scale (DAS-18B) from baseline to post-assessment (t0 to t1) and follow-up (t0 to t2); 18 items are assessed on a 7-point Likert scale; high score indicates more dysfunctional beliefs (minimum = 18; maximum = 126)
Mental Well-Being (Warwick-Edinburgh Mental Well-being Scale) | baseline (t0), post (10 weeks; t1), and follow-up (3 months; t2)
  Change in mental well-being as measured by the short version of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) from baseline to post-assessment (t0 to t1) and follow-up (t0 to t2); 14 items assessed on a 5-point Likert scale (minimum = 14; maximum = 70). Higher scores indicate better well-being.
Resilience (Resilience Scale) | baseline (t0), post (10 weeks; t1), and follow-up (3 months; t2)
  Change in resilience as measured by the 13-item Resilience Scale from baseline to post-assessment (t0 to t1) and follow-up (t0 to t2); 13 items assessed on a 7-point Likert scale (minimum = 13; maximum = 91). Higher scores indicate more resilience.
Rumination (Ruminative Responses Scale) | baseline (t0), post (10 weeks; t1), and follow-up (3 months; t2)
  Change in rumination measured by the Ruminative Response Scale (RRS) from baseline to post-assessment (t0 to t1) and follow-up (t0 to t2); 10 items assessed on a 4-point Likert scale (minimum = 10; maximum = 40). Higher scores indicate more ruminative behaviors.
Loneliness (UCLA Loneliness scale) | baseline (t0), post (10 weeks; t1), and follow-up (3 months; t2)
  Change in loneliness as measured by the 3-item UCLA Loneliness scale from baseline to post-assessment (t0 to t1) and follow-up (t0 to t2); 3-items assessed on a 4-point Likert scale (minimum = 4; maximum = 12). Higher scores indicate more loneliness.
Self-rated health (EQ5D5L Visual Analog Scale ) | baseline (t0), post (10 weeks; t1), and follow-up (3 months; t2)
  Change in self-rated health as measured by the EQ5D5L Visual Analog Scale from baseline to post-assessment (t0 to t1) and follow-up (t0 to t2); Rating Scale 0 (worst health possible) - 100 (best health possible).
Session-specific effects | Before and after each session weeks 1 through 10
  Before and after each session during weeks 1 through 10, participants will complete a 40-item questionnaire regarding changes in depressive symptoms, negative (meta)cognitive beliefs and attitudes associated with depression, which are targeted in the MCT-Silver BeWell. Items are assessed on a 6-point LIkert scale (minimum = 40; maximum = 240); high scores indicate more negative beliefs / attitudes

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Viertel, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moritz S, Menon M, Balzan R, Woodward TS. Metacognitive training for psychosis (MCT): past, present, and future. Eur Arch Psychiatry Clin Neurosci. 2023 Jun;273(4):811-817. doi: 10.1007/s00406-022-01394-9. Epub 2022 Mar 25. PMID 35338378
- [Background] Miegel F, Rubel J, Dietrichkeit M, Hagemann-Goebel M, Yassari AH, Balzar A, Scheunemann J, Jelinek L. Exploring mechanisms of change in the metacognitive training for depression. Eur Arch Psychiatry Clin Neurosci. 2024 Apr;274(3):739-753. doi: 10.1007/s00406-023-01604-y. Epub 2023 Apr 17. PMID 37067579
- [Background] Jelinek L, Hauschildt M, Wittekind CE, Schneider BC, Kriston L, Moritz S. Efficacy of Metacognitive Training for Depression: A Randomized Controlled Trial. Psychother Psychosom. 2016;85(4):231-4. doi: 10.1159/000443699. Epub 2016 May 27. No abstract available. PMID 27230865
- [Background] Wu JJ, Wang HX, Yao W, Yan Z, Pei JJ. Late-life depression and the risk of dementia in 14 countries: a 10-year follow-up study from the Survey of Health, Ageing and Retirement in Europe. J Affect Disord. 2020 Sep 1;274:671-677. doi: 10.1016/j.jad.2020.05.059. Epub 2020 May 26. PMID 32664001
- [Background] Yip PSF, Zheng Y, Wong C. Demographic and epidemiological decomposition analysis of global changes in suicide rates and numbers over the period 1990-2019. Inj Prev. 2022 Apr;28(2):117-124. doi: 10.1136/injuryprev-2021-044263. Epub 2021 Aug 16. PMID 34400542
- [Background] Schaakxs R, Comijs HC, Lamers F, Kok RM, Beekman ATF, Penninx BWJH. Associations between age and the course of major depressive disorder: a 2-year longitudinal cohort study. Lancet Psychiatry. 2018 Jul;5(7):581-590. doi: 10.1016/S2215-0366(18)30166-4. Epub 2018 Jun 18. PMID 29887519
- [Background] Reynolds CF 3rd, Jeste DV, Sachdev PS, Blazer DG. Mental health care for older adults: recent advances and new directions in clinical practice and research. World Psychiatry. 2022 Oct;21(3):336-363. doi: 10.1002/wps.20996. PMID 36073714
- [Background] Schneider BC, Veckenstedt R, Karamatskos E, Ahlf-Schumacher J, Gehlenborg J, Schultz J, Moritz S, Jelinek L. Efficacy and moderators of metacognitive training for depression in older adults (MCT-Silver): A randomized controlled trial. J Affect Disord. 2024 Jan 15;345:320-334. doi: 10.1016/j.jad.2023.10.118. Epub 2023 Oct 19. PMID 37865342
- [Background] Schneider BC, Bücker L, Riker S, Karamatskos E, Jelinek L. A pilot study of metacognitive training (D-MCT) for older adults with depression. Zeitschrift für Neuropsychologie. 2018; 29.
- [Background] Volz HP, Stirnweiss J, Kasper S, Moller HJ, Seifritz E. Subthreshold depression - concept, operationalisation and epidemiological data. A scoping review. Int J Psychiatry Clin Pract. 2023 Mar;27(1):92-106. doi: 10.1080/13651501.2022.2087530. Epub 2022 Jun 23. PMID 35736807
- [Background] Hauschildt M, Arlt S, Moritz S, Yassari AH, Jelinek L. Efficacy of metacognitive training for depression as add-on intervention for patients with depression in acute intensive psychiatric inpatient care: A randomized controlled trial. Clin Psychol Psychother. 2022 Sep;29(5):1542-1555. doi: 10.1002/cpp.2733. Epub 2022 Mar 21. PMID 35274407